CLINICAL TRIAL: NCT03077074
Title: Brain Responses to Visual Food Cues in Response to a Low Carbohydrate Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ram Weiss, Ram Weiss, clinical professor and principle investigator, Hadassah Medical Organization
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 12-0580-HMO
Record Dates: First submitted 2017-02-20; First posted 2017-03-10 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Changes in Functional MRI

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low carbohydrate consumption (Experimental): consumption of up to 60 grams of carbohydrate a day for 10 days FMRI will be performed prior and after the intervention during the luteal cycle phase
  Interventions: Other: low carbohydrate consumption

INTERVENTIONS:
Other: low carbohydrate consumption — consumption of up to 60 grams of carbohydrate a day for 10 days FMRI will be performed prior and after the intervention during the luteal cycle phase

SUMMARY:
The aim is to profile and elucidate the hormonal and neurological system interaction to food related behavior. The stimulus used will include visual and taste (gustatory) stimuli. The study will profile induced correlations of metabolic parameters, gut hormones and brain region (ROI - regions of interest) activation and interaction. In this study we will use fMRI (functional MRI) to compare brain responses in obese, normal-weight and reduced weight subjects. The food stimuli will be blocked into specific categories to allow for investigation of different responses to alternating energy density foods. The response will be tested prior to and following a brief low carbohydrate dietary regimen.

DETAILED DESCRIPTION:
The study will be a longitudinal study where the participants will come back twice on the same phase of the period- both visits in the luteal phase with a month between each visit. In this part of the study there will be 40 participants with a wider range of BMI. This phase of the study will include a nutritional intervention - the participants will be asked to have a carbohydrate restricted diet (60 grams of carbohydrate)- for a period of a month with no caloric restriction. Food records will be kept and followed and a ketone test (blood test) will be done on the morning of the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 45 years
* No contraindication to enter the MRI
* No significant visual problems that may hamper visualization of visual stimuli within the magnet
* No contraceptive hormonal replacement
* relatively regular menstrual cycle

Exclusion Criteria:

* contraceptive hormonal replacement
* under the age of 18
* over the age of 45
* pharmacological treatment that can effect brain response
* Irregular menstrual cycle

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females without contraceptive treatment and with regular menstrual cycle
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
fMRI:(Functional MRI) changes in activation patterns of reward associated regions will be assessed prior and after dietary intervention | fMRI will be preformed in the luteal menstrual phase at two time points (at least a month apart). a comparison will be made between pre and post intervention.
  BOLD (Blood Oxygen Level Dependent) responses will we quantified in regions of interest

CONTACTS AND LOCATIONS:
Overall Officials: Ram Weiss, Professor, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah hebrew university, Jerusalem Region, Israel

IPD SHARING:
Plan to Share IPD: No